CLINICAL TRIAL: NCT07267962
Title: The Effect of ChatGPT-5, Gemini 2.5 Pro, and DeepSeek V3.1 Guided Rehabilitation on Clinical Outcomes in Individuals With Degenerative Knee Disease
Brief Title: LLM-Guided Rehabilitation in Degenerative Knee Disease
Acronym: LLM-RehabKnee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Omer Alperen Gurses, Ph.D. Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025/1056
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Knee Disease
Keywords: Degenerative knee disease; physiotherapy; rehabilitation; large language model; ChatGPT; DeepSeek; Gemini

STUDY DESIGN:
Intervention Model Description: Four-arm, parallel-group randomized controlled trial in adults with degenerative knee disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional physiotherapy (Active Comparator): Participants receive supervised conventional physiotherapy including hot pack, TENS, ultrasound and a standardized knee exercise program two times per week for 8 weeks (16 sessions).
  Interventions: Biological: Supervised conventional physiotherapy
- Conventional physiotherapy plus ChatGPT-5-assisted exercise planning (Experimental): Participants receive supervised conventional physiotherapy plus an exercise program whose content and progression are planned with the assistance of the ChatGPT-5 large language model, under physiotherapist supervision, two times per week for 8 weeks (16 sessions).
  Interventions: Behavioral: ChatGPT-5-assisted exercise planning
- Conventional physiotherapy plus DeepSeek V3.1-assisted exercise planning (Experimental): Participants receive supervised conventional physiotherapy plus an exercise program whose content and progression are planned with the assistance of the DeepSeek V3.1 large language model, under physiotherapist supervision, two times per week for 8 weeks (16 sessions).
  Interventions: Behavioral: DeepSeek V3.1-assisted exercise planning
- Conventional physiotherapy plus Gemini 2.5 Pro-assisted exercise planning (Experimental): Participants receive supervised conventional physiotherapy plus an exercise program whose content and progression are planned with the assistance of the Gemini 2.5 Pro large language model, under physiotherapist supervision, two times per week for 8 weeks (16 sessions).
  Interventions: Behavioral: Gemini 2.5 Pro-assisted exercise planning

INTERVENTIONS:
Biological: Supervised conventional physiotherapy — Supervised outpatient physiotherapy including hot pack (20 minutes), conventional TENS (100 Hz, 60 µs, 20 minutes), therapeutic ultrasound (1 MHz, 1.5 W/cm², 5 minutes) and a standardized knee exercise program (strengthening, range of motion, proprioceptive and functional exercises), delivered two times per week for 8 weeks (16 sessions in total).
  Arms: Conventional physiotherapy
Behavioral: ChatGPT-5-assisted exercise planning — Exercise selection and progression for the knee rehabilitation program supported by standardized prompts to the ChatGPT-5 large language model. All LLM-generated suggestions are reviewed for safety and appropriateness by physiotherapists before being implemented in supervised sessions.
  Arms: Conventional physiotherapy plus ChatGPT-5-assisted exercise planning
Behavioral: DeepSeek V3.1-assisted exercise planning — Exercise selection and progression for the knee rehabilitation program supported by standardized prompts to the DeepSeek V3.1 large language model. All LLM-generated suggestions are reviewed for safety and appropriateness by physiotherapists before being implemented in supervised sessions.
  Arms: Conventional physiotherapy plus DeepSeek V3.1-assisted exercise planning
Behavioral: Gemini 2.5 Pro-assisted exercise planning — Exercise selection and progression for the knee rehabilitation program supported by standardized prompts to the Gemini 2.5 Pro large language model. All LLM-generated suggestions are reviewed for safety and appropriateness by physiotherapists before being implemented in supervised sessions.
  Arms: Conventional physiotherapy plus Gemini 2.5 Pro-assisted exercise planning

SUMMARY:
This randomized, four-arm clinical trial will investigate the effects of large language model (LLM)-assisted exercise prescriptions integrated with conventional physiotherapy on pain, function and quality of life in adults with degenerative knee disease. Participants will be randomly assigned to conventional physiotherapy alone or to conventional physiotherapy plus an exercise program planned with the assistance of ChatGPT-5, Gemini 2.5 Pro, or DeepSeek V3.1. All participants will receive supervised outpatient physiotherapy two times per week for 8 weeks (16 sessions in total). Outcomes will be assessed at baseline and at the end of the 8-week intervention period by physiotherapists blinded to group allocation.

DETAILED DESCRIPTION:
Degenerative knee disease, including knee osteoarthritis, is a common cause of pain, disability and loss of independence in middle-aged and older adults. Exercise-based rehabilitation is a core component of evidence-based management, but the content and progression of exercise programs often vary between clinicians. Large language models (LLMs) such as ChatGPT-5, DeepSeek V3.1 and Gemini 2.5 Pro can generate exercise suggestions based on clinical information and may support physiotherapists in designing and progressing individualized programs. However, their impact on clinical outcomes in degenerative knee disease has not been evaluated in randomized controlled trials.

This single-center, randomized, parallel-group clinical trial will be conducted in adults with degenerative knee disease referred to the physiotherapy clinic of Kirsehir Ahi Evran University. After written informed consent and baseline assessments, participants will be randomly assigned (1:1:1:1) to one of four groups. All groups will receive a standardized outpatient physiotherapy program including hot pack, conventional TENS, therapeutic ultrasound and strengthening, range of motion, proprioceptive and functional exercises for the knee joint. In the three experimental groups, the content and progression of the exercise program will be planned with the assistance of standardized prompts to ChatGPT-5, DeepSeek V3.1 or Gemini 2.5 Pro, and all LLM-generated suggestions will be reviewed for safety and appropriateness by physiotherapists before being implemented. Sessions will be delivered two times per week for 8 weeks (16 supervised visits) under the supervision of a physical medicine and rehabilitation specialist and physiotherapists.

Outcomes will be evaluated at baseline (week 0) and after the 8-week intervention by a physiotherapist blinded to group allocation. Main outcome domains include knee pain, knee-related patient-reported outcomes, objective functional performance tests, isometric muscle strength, knee range of motion, psychosocial factors and health-related quality of life. Data will be analyzed according to CONSORT guidelines for randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years.
* Clinical and radiographic diagnosis of degenerative knee disease in the target knee.
* Knee pain in the target knee for at least 3 months.
* Ability to bear weight on the target limb and perform the planned functional tests.
* Sufficient cognitive and physical capacity to participate in an 8-week supervised exercise program.
* Willingness to participate and ability to provide written informed consent.

Exclusion Criteria:

* Intra-articular corticosteroid or similar injection to the target knee within the previous 3 months.
* Knee surgery on the target knee within the previous 6 months.
* Severe malalignment of the knee or concomitant severe neurological disease and/or balance disorder that would interfere with safe testing or exercise.
* Pregnancy or any systemic disease that would contraindicate participation in the rehabilitation program according to the physician.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in WOMAC total score | Baseline (week 0) to end of treatment (week 8)
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score (0-96), composed of pain, stiffness and physical function subscales. Higher scores indicate worse symptoms and function. The primary analysis will compare change in WOMAC total score from baseline to week 8 between the four groups.

SECONDARY OUTCOMES:
Change in knee pain intensity at rest, at night and during activity (Numeric Pain Rating Scale) | Baseline (week 0) to week 8
  Numeric Pain Rating Scale (0-10) scores for knee pain at rest, at night and during activity. Higher scores indicate more severe pain. Mean change in each pain condition from baseline to week 8 will be compared between groups.
Change in IKDC subjective knee score | Baseline (week 0) to week 8
  International Knee Documentation Committee (IKDC) subjective knee form score (0-100). Higher scores indicate better symptoms, sports activity and knee function. Change from baseline to week 8 will be compared between groups.
Change in Lysholm knee score | Baseline (week 0) to week 8
  Lysholm knee score (0-100). Higher scores indicate better knee function. Change from baseline to week 8 will be analyzed between the four groups.
Change in 30-second chair stand test performance | Baseline (week 0) to week 8
  Number of full stands completed in 30 seconds from a standard chair. Higher numbers indicate better lower limb functional performance. Change in repetitions from baseline to week 8 will be compared between groups.
Change in fast walking test time | Baseline (week 0) to week 8
  Time (seconds) required to complete a fast walking test over a fixed distance (e.g., 4 × 10 m or 40 m, according to the study protocol). Lower times indicate better performance. Change in time from baseline to week 8 will be analyzed.
Change in stair climb test time | Baseline (week 0) to week 8
  Time (seconds) needed to ascend and/or descend a standardized set of stairs. Lower times indicate better functional performance. Change from baseline to week 8 will be compared between groups.
Change in maximal isometric quadriceps strength | Baseline (week 0) to week 8
  Maximal voluntary isometric strength of the quadriceps muscle of the target knee, measured with a handheld dynamometer. Higher values (e.g., Newtons) indicate greater muscle strength. Change from baseline to week 8 will be compared between groups.
Change in maximal isometric hamstring strength | Baseline (week 0) to week 8
  Maximal voluntary isometric strength of the hamstring muscles of the target limb, measured with a handheld dynamometer. Higher values indicate greater muscle strength. Change from baseline to week 8 will be compared between groups.
Change in knee range of motion | Baseline (week 0) to week 8
  Active knee flexion and extension range of motion measured with a universal goniometer in degrees. Higher flexion and closer-to-zero extension deficit indicate better joint mobility. Changes in range of motion from baseline to week 8 will be analyzed.
Change in Pain Catastrophizing Scale score | Baseline (week 0) to week 8
  Pain Catastrophizing Scale total score (0-52). Higher scores indicate greater levels of pain catastrophizing. Change from baseline to week 8 will be compared between groups.
Change in Tampa Scale for Kinesiophobia score | Baseline (week 0) to week 8
  Tampa Scale for Kinesiophobia total score (17-68). Higher scores indicate greater fear of movement or re-injury. Change from baseline to week 8 will be analyzed between groups.
Change in Hospital Anxiety and Depression Scale - Anxiety subscale score | Baseline (week 0) to week 8
  Hospital Anxiety and Depression Scale (HADS) - Anxiety subscale score (0-21). Higher scores indicate higher anxiety symptoms. Change from baseline to week 8 will be compared between groups.
Change in Hospital Anxiety and Depression Scale - Depression subscale score | Baseline (week 0) to week 8
  Hospital Anxiety and Depression Scale (HADS) - Depression subscale score (0-21). Higher scores indicate higher depressive symptoms. Change from baseline to week 8 will be analyzed between groups.
Change in SF-12 physical and mental component summary scores | Baseline (week 0) to week 8
  Short Form-12 (SF-12) physical and mental component summary scores (0-100). Higher scores indicate better health-related quality of life. Change from baseline to week 8 will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Merez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because there is currently no approved institutional or ethical framework for external IPD sharing in this study.